CLINICAL TRIAL: NCT01627431
Title: Tailored Strategy for Residual Platelet Activity In Advanced Peripheral Artery Disease: New Optimal Management.
Brief Title: Residual Platelet Activity In Advanced Peripheral Artery Disease
Acronym: TRAIANO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Francesco Violi, Prof., University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SAPIENZA-PAD
Record Dates: First submitted 2012-06-14; First posted 2012-06-25 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Peripheral revascularization; Antiplatelet therapy; Residual platelet activity
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antiplatelet therapy (Other): Patients underwent peripheral revascularization procedures undergoing a double antiplatelet therapy
  Interventions: Drug: Acetylsalicylic acid; Drug: Clopidogrel

INTERVENTIONS:
Drug: Acetylsalicylic acid — 100 mg once per day
  Other Names: Aspirin
Drug: Clopidogrel — 75 mg once per day
  Other Names: Plavix

SUMMARY:
The peripheral arterial disease (PAD) is a common atherosclerotic disease manifestation and its prevalence increase with age and with the simultaneous presence of cardiovascular risk factors.

PAD patients are usually treated, as a first line treatment, with the exercise therapy, combined with the pharmacological antiplatelet therapy.

In the case of first line therapy failure, PAD patients usually undergoing to invasive revascularization procedures.

After a peripheral stent has been located, the major follow-up problem is the restenosis rate.

Published studies describe how, in a large amount of patients, can be recognised an high residual platelet activity. These data about PAD patients at the moment are lacking .

The authors would evaluate the incidence of PAD patients with an high residual platelet activity.

DETAILED DESCRIPTION:
The peripheral arterial disease (PAD) is a common atherosclerotic disease manifestation and its prevalence increases with age and with the co-presence of cardiovascular risk factors. PAD affects a large proportion of the adult population, with an age-adjusted prevalence of 4-15% which increases to 29% in case of comorbidity such as the presence of diabetes mellitus in the same individual. Less than 20% of patients with peripheral arterial laments the typical symptom of "claudication intermittens". Studies on the symptomatic PAD natural history indicate that the risk of limb loss in non-diabetic patients is low (2% or less), but the cardiovascular disease represent the leading cause of death; the annual rate of cardiovascular events (myocardial infarction, stroke or cardiovascular death) is between 5 and 7%. Medical treatment and / or surgery in this type of patient should be directed not only to improve the walking autonomy but also to reduce cardiovascular risk. Claudicant patients first-line therapy is based on structured physical exercise program and, in some specific cases, on the antiplatelet pharmacological therapy. The lack of response to exercise and / or drug therapy should lead to the next level of decision making, which is to consider limb revascularization procedures. However, in patients with suspected proximal lesion (gluteal claudication or absent femoral pulse), revascularization procedures could be considered as a first line therapy. When the revascularization procedures are considered, the first choice intervention should be the endovascular strategy, considering the lowest number of periprocedural complications. Recommendations for optimal drug therapy after revascularisation procedures in the lower limbs are hampered by lack of agreement on the optimal role of these procedures, and lack of data from randomized clinical trials. Transluminal angioplasty (PTA), primary or associated with stenting, is recommended for focal stenotic lesions of the iliac (common and external first section) and femoral-popliteal axis, particularly when the claudication intermittents is considered as severe, rather than critical ischemia. Also, this approach is recommended in non-diabetic patients with a relatively preserved tibial vessels flow. Exists a minor agreement about endovascular procedures use in extended occlusive lesions. In recent years, has become more common the use of open or covered stents during endovascular treatments in order to make it more secure and durable over time, especially in obstructive and extended lesions. This has certainly led to improved primary patency outcomes, but has entailed and still entails additional problems of drug therapy agreement.

Nowadays, the main problem concerning lower limbs revascularization is the post-procedure anti-thrombotic pharmacological treatment and the different antiplatelet drugs effectiveness This issue was addressed in two meta-analyses, where have been shown how the data are not conclusive. Moreover, a recent study by Marcucci et al (Circulation. 2009; 119: 237-42) has clearly shown that impaired platelet activation inhibition is a crucial point for the prevention of vascular outcomes, because residual platelet reactivity has been associated with adverse vascular outcomes.

Overall, these data identify two key issues:

1. Platelet hyperactivation, usually observed after revascularization procedures;
2. The platelet inhibition percentage appears crucial to reduce postoperative thrombotic complications and restenosis early onset.

Therefore, a unique aspect of this study is to analyze whether after peripheral revascularization procedures a platelet hyperactivation is observed and evaluate the possible involved mechanisms. In fact, the knowledge of the underlying mechanism could lead to more appropriate pharmacological approach to prevent platelet activation. In this context, the authors would explore the role of reactive oxygen species (ROS) in inducing platelet activation in patients with PAD undergoing revascularization devices.

ELIGIBILITY:
Inclusion Criteria:

* Claudicatio Intermittens affected patients in which both exercise than pharmacological therapies failed
* Ankle Brachial Index < 0.9 or > 1.3
* Peripheral Arteries stenosis > 50% bilateral

Exclusion Criteria:

* Acute Limb Ischemia patients
* Patients that underwent a peripheral revascularization procedure within 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Residual Platelet Activity | 2 years
  Evaluate the high residual platelet activity prevalence in PAD patients

SECONDARY OUTCOMES:
Target vessels thrombosis | 2 years
  Evaluate the target vessels thrombosis incidence
Major Cardiac Events | 2 years
  Evaluate the Major Cardiac Events (MACE) incidence in PAD patients undergoing the peripheral revascularization procedures.
Platelet aggregation tests | 2 years
  Compare the different platelet aggregation tests specificity, sensitivity, accuracy and predictive values
Oxidative stress | 2 years
  Evaluate platelet activation and oxidative stress indexes relationship
Laboratory tests predictive values | 2 years
  Evaluate the different laboratory tests (platelet aggregation, oxidative stress markers, seric thromboxane) predictive values in identify recurrent thrombosis high risk patients
High risk patients score | 2 years
  Validate a clinical-laboratoristic predictive score in order to identify recurrent thrombosis high risk patients

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — Divisione di Prima Clinica Medica - Sapienza University of Rome; Rosanna Abate, MD, Study Chair — Azienda Ospedaliero-Universitaria Careggi University of Florence
Locations (2):
- Italy (2):
  - University of Florence - Azienda Ospedaliero-Universitaria Careggi, Florence, Florence
  - Sapienza- University of Rome -Azienda Policlinico Umberto I, Rome, Rome